CLINICAL TRIAL: NCT00513916
Title: Effects of Soy on Estrogens in Breast Fluid and Urine
Brief Title: Effect of Dietary Soy on Estrogens in Breast Fluid, Blood, and Urine Samples From Healthy Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Hawaii Cancer Research Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Gertraud Maskarinec, Cancer Research Center of Hawaii
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: CDR0000560821; UHM-CHS-4116
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2009-04

CONDITIONS: Breast Cancer; Healthy, no Evidence of Disease
Keywords: breast cancer; healthy, no evidence of disease
MeSH Terms: conditions — Breast Neoplasms | interventions — Soybean Proteins

ARMS (2):
- Arm I (Experimental): Participants partake in a high soy diet consisting of 2 daily soy servings (approximately 50mg isoflavones).
  The choice of soy foods will include ½ cup of tofu, ¾ cup of soy milk, or ¼ cup of soy nuts. Replacement of currently consumed foods with soy foods will be encouraged.
  Interventions: Dietary Supplement: soy isoflavones
- Arm II (Active Comparator): Participants will be asked to keep their soy intake below 3 servings per week. The participants will also receive general nutrition counseling.
  Interventions: Dietary Supplement: soy isoflavones

INTERVENTIONS:
Dietary Supplement: soy isoflavones — High or low dose of soy isoflavones in the diet.

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. Eating a diet high in isoflavones, compounds found in soy foods, may keep cancer from forming.

PURPOSE: This randomized phase III trial is studying the effects of dietary soy on estrogens in breast fluid, blood, and urine samples from healthy women.

DETAILED DESCRIPTION:
OBJECTIVES:

* Examine the effects of two daily servings of soy on estrogen levels in nipple aspirate fluid (NAF) and serum.
* Investigate cytologic patterns of epithelial breast cells obtained from NAF as a measure of proliferation in relation to soy intake.
* Explore the effect of two daily servings of soy on cytochrome alterations of estrogen metabolism as expressed in the formation of urinary 2-, 16α-, and 4-hydroxy estrogen metabolites.
* Compare estrogen levels in NAF and serum measured at the same time during the luteal phase.

OUTLINE: This is a multicenter study. Participants are randomized to 1 of 2 intervention arms.

* Arm I: Participants partake in a high soy diet consisting of 2 daily soy servings (approximately 50mg isoflavones). The choice of soy foods will include ½ cup of tofu, ¾ cup of soy milk, or ¼ cup of soy nuts. Replacement of currently consumed foods with soy foods will be encouraged.
* Arm II: Participants will be asked to keep their soy intake below 3 servings per week. The participants will also receive general nutrition counseling.

In both arms, intervention continues for 6 months. After 6 months, participants undergo a 1-month washout period and then cross-over to the other intervention arm.

Nipple aspirate fluid, urine, and blood samples are collected periodically to measure laboratory endpoints.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy participant

  * No diagnosis of cancer

PATIENT CHARACTERISTICS:

* Premenopausal
* Regular menstrual cycles

PRIOR CONCURRENT THERAPY:

* Not taking birth control pills or other hormones

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-07; Primary Completion 2011-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Effect of two daily servings of soy on estrogen levels in nipple aspirate fluid (NAF) and serum
Cytologic patterns of epithelial breast cells obtained from NAF
Effect of two daily servings of soy on cytochrome alterations of estrogen metabolism as expressed in the formation of urinary 2-, 16α-, and 4-hydroxy estrogen metabolites
Comparison of estrogen levels in NAF and serum measured at the same time during luteal phase

CONTACTS AND LOCATIONS:
Overall Officials: Gertraud Maskarinec, MD, PhD, Study Chair — University of Hawaii Cancer Research Center
Locations (1):
- Cancer Research Center of Hawaii, Honolulu, Hawaii, United States

REFERENCES:
- [Result] Sen C, Morimoto Y, Heak S, Cooney RV, Franke AA, Maskarinec G. Soy foods and urinary isoprostanes: results from a randomized study in premenopausal women. Food Funct. 2012 May;3(5):517-21. doi: 10.1039/c2fo10251j. Epub 2012 Feb 14. PMID 22331037
- [Result] Maskarinec G, Morimoto Y, Conroy SM, Pagano IS, Franke AA. The volume of nipple aspirate fluid is not affected by 6 months of treatment with soy foods in premenopausal women. J Nutr. 2011 Apr 1;141(4):626-30. doi: 10.3945/jn.110.133769. Epub 2011 Feb 16. PMID 21325473
- [Derived] Maskarinec G, Suzuki S, Pagano IS, Morimoto Y, Franke AA, Ehya H. Cytology in nipple aspirate fluid during a randomized soy food intervention among premenopausal women. Nutr Cancer. 2013;65(8):1116-21. doi: 10.1080/01635581.2013.833638. Epub 2013 Oct 15. PMID 24127645